CLINICAL TRIAL: NCT07104877
Title: A Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of SYH2051 in Combination With SYS6010 in Patients With Gastrointestinal Tumors Such as Advanced Colorectal Cancer
Brief Title: A Study of SYS6010 in Combination With SYH2051 in Patients With Advanced Colorectal Cancer and Other Gastrointestinal Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYH2051-002
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Gastric Cancer (GC); Gastrointestinal Tumors
Keywords: SYS6010; SYH2051
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYS6010+SYH2051 (Experimental)
  Interventions: Drug: SYS6010; Drug: SYH2051

INTERVENTIONS:
Drug: SYS6010 — Administered via intravenous infusion at the dose of 3.2-4.8 mg/kg
Drug: SYH2051 — Administered via oral at the dose of 40-80 mg

SUMMARY:
This study is an open-label, non-randomized trial design, including a dose escalation phase and a dose expansion phase, to evaluate the safety, tolerability and preliminary anti-tumor activity of SYS6010 in combination with SYH2051 in patients with advanced gastrointestinal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients with unresectable or metastatic colorectal cancer or other gastrointestinal tumors confirmed by histology or pathology, who have failed at least first-line standard therapy or for whom standard treatment is not applicable.
* Provide tumor tissue samples for immunohistochemical EGFR expression testing, with EGFR expression positive as confirmed by the central laboratory.
* At least one measurable lesion confirmed according to RECIST v 1.1 criteria.
* ECOG performance status score of 0-1.
* Expected survival of ≥3 months.
* Major organ functions must meet relevant laboratory criteria for blood counts, renal function, liver function, and coagulation within 7 days prior to treatment.
* Subjects agree to use effective contraception during the study and for 6 months after the last dose, with women being non-lactating and men refraining from sperm donation. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first administration of the study drug.
* Willing to participate in the study, understand the study procedures, and sign a written informed consent form.

Exclusion Criteria:

* Previously treated with antibody-drug conjugates (ADC) containing topoisomerase I inhibitors.
* Failure to meet the required washout period for prior medications or treatments as specified in the protocol..
* Has other primary malignancies within 3 years prior to the first dose of the study drugs.
* History of severe cardio-cerebrovascular disease.
* Adverse events from prior anti-tumor treatments that have not resolved to ≤ Grade 1 of CTCAE V5.0.
* Patients with active central nervous system and/or leptomeningeal metastases.
* Clinically significant pleural effusion, peritoneal effusion, or pericardial effusion requiring intervention.
* Has a history of Interstitial lung disease (ILD)/non-infectious pneumonitis that required steroids, has current ILD/non-infectious pneumonitis, or where suspected ILD/non-infectious pneumonitis cannot be ruled out by imaging at screening.
* Patients with thyroid dysfunction requiring treatment, but that well-controlled was allowed.
* Severe infections within 4 weeks prior to the first administration of the study drugs.
* Prior interruption of EGFR-targeted therapy due to skin toxicity, or skin diseases requiring oral or intravenous treatment currently.
* Known allergy to any component of SYS6010 or SYH2051, or any humanized monoclonal antibody product.
* Severe ophthalmic history (e.g., dry eye syndrome, keratitis, conjunctivitis, etc.).
* Had a history of autoimmune disease (except tuberous sclerosis), immunodeficiency (including positive HIV test), or other acquired or congenital immunodeficiency diseases, or organ transplantation.
* Active HBV, HCV infection or syphilis infection.
* Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Up to 90 days following the last dose
  Occurrence and frequency of Adverse Event (AE)The occurrence and incidence of adverse events (AEs) will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. AEs will be monitored from the first dose until the safety follow-up period.
Dose-limiting toxicities (DLTs) | Up to 21 days
  DLTs are defined as adverse events related to the study drug that meet the protocol-specified criteria for dose limitation.

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 | Up to 2 years
  The objective response rate (ORR) will be assessed based on RECIST v1.1 criteria. ORR is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) as the best overall response.
Disease Control Rate (DCR) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Progression-free Survival (PFS) | Up to 2 years
Overall survival (OS) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Cancer Hospital, Fuzhou, Fujian, China